CLINICAL TRIAL: NCT01212679
Title: Pilot Study of Intranasal Nerve Growth Factor for Traumatic Brain Injury(TBI)
Brief Title: Effects of Intranasal Nerve Growth Factor for Traumatic Brain Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Xinfeng Liu, Professor, Jinling Hospital, China
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGF-TBI
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2016-11

CONDITIONS: Traumatic Brain Injury
Keywords: nerve growth factor; traumatic brain injury; intranasal; prognosis; neurological function
MeSH Terms: conditions — Brain Injuries, Traumatic; Hereditary Sensory and Autonomic Neuropathies | interventions — Nerve Growth Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nerve growth factor (Experimental): Patients who underwent TBI will be chosen to receive NGF randomly.
  Interventions: Drug: nerve growth factor
- Control (Placebo Comparator): Patients who underwent TBI will be chosen to receive nomral saline randomly.
  Interventions: Drug: nomral saline

INTERVENTIONS:
Drug: nerve growth factor — The experimental group patients will receive NGF 20ug/d intranasally for 2 weeks.
  Arms: nerve growth factor
Drug: nomral saline — The Placebo Comparator group patients will receive nomral saline 20ug/d intranasally for 2 weeks.
  Arms: Control

SUMMARY:
Traumatic bain injury(TBI) remains a hidden epidemic involving individuals affected predominantly at a young age who in the most severe cases remain with permanent physical,psychological and cognitive deficits.This study will investigate the therapeutic effects of intranasal Nerve Growth Factor(NGF) in TBI.

DETAILED DESCRIPTION:
Early NGF concentration in the cerebral spinal fluid(CSF)correlates significantly with the severity of head injury, and NGF upregulation correlates with better neurologic outcomes and could be useful to obtain clinical and prognostic information in patients with serve TBI.

However, the clinical use of NGF is difficulty associated with delivering them to the CNS because of the existing of blood-brain barrier(BBB). Intranasal delivery drug is a noninvasive and convenient novel method bypassing BBB, which results in targeting therapeutics to the CNS rapidly.

The proposed study is a randomized, double-blind, placebo-controlled trail of NGF, starting between 24 to 72 hours post TBI, continuing for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

Moderate to severe blunt traumatic brain injury defined as Glasgow Coma Scale(GCS) between 7 and 13.

Age 18~65 years. Admission to Jinling Hospital between 24 to 72 hours. Subjects capable of giving informed consent or have an acceptable surrogate capable of giving consent on the subject's behalf.

Exclusion Criteria:

Skull fracture, Cerebrospinal fluid rhinorrhea. Severe concurrent illness with life expectancy<6 months or other serious illness which have a major impact on the outcome.

Treatment with other investigational agents in the past 4 weeks. Allergy to NGF. Primary ciliary dyskinesia, Asthma, Cystic fibrosis, Viral and bacterial infections, Diabetes mellitus.

Inability to provide informed consent. Pregnancy or breast-breeding. Women of childbearing age will be given a pregnancy test during screening to exclude pregnancy.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2010-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
improved neurological functions | at months 6 post-treatment
  Neurological functions will be assessed by GOS(Glasgow Outcome Scale), mRS(modified Rankin Scale),BI(Barthel index).

SECONDARY OUTCOMES:
HAMA,HAMD | at months 6 post-treatment
  HAMA(Hamilton Anxiety Scale ),HAMD(Hamilton Depression Scale).

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, MD, Study Chair — Department of Neurology, Jinling Hospital, Nanjing University School of Medicine
Locations (1):
- Department of Neurology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided